CLINICAL TRIAL: NCT06228846
Title: An Open-Label Phase I Study to Evaluate the Safety,Tolerability and Preliminary Efficacy of YY001 in Patients with Advanced Solid Tumors
Brief Title: An Phase I Study of YY001 in Patients with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yuyao Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-YY001-CH1
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study treatment (Experimental): Method of Administration: Single dose period: Single oral ; Multiple dose period: Oral , QD.
  Interventions: Drug: YY001

INTERVENTIONS:
Drug: YY001 — Oral

SUMMARY:
The safety and tolerability of YY001 in the treatment of patients with advanced solid tumors were evaluated, and the possible dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD) or recommended phase II clinical dose (RP2D) were observed.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients fully understand and sign ICF, voluntarily participate in the study, and able to follow and complete all study procedures.
* 2. Aged 18-75 years (including upper and lower limits), male or female.
* 3. Patients with histologically or cytologically confirmed advanced unresectable or metastatic solid tumors (mainly gastrointestinal tumors such as colorectal cancer and gastric cancer, and prostate cancer)
* 4.The standard treatment failure (disease progression after treatment or treatment side effects not tolerance), or top treatment, or shall not apply to the current standard treatment for patients
* 5. For patients with advanced solid tumors (dose-escalation phase), at least one tumor lesion that could be evaluated according to RECIST, version 1.1; (Dose-expansion phase) At least one measurable tumor lesion according to RECIST, version 1.1 (a tumor that is located in the previously irradiated area or another locoregional treatment site and is generally not considered a measurable lesion unless there is definite progression or persistence beyond 3 months of radiation);
* 6. ECOG physical condition≤1
* 7. Patients with advanced primary liver cancer should meet the Child-Pugh liver function grading: grade A and better grade B (≤7).
* 8. With adequate bone marrow, liver and kidney organ function:

  •Blood system within 14 days (not received blood transfusions or hematopoietic stimulating factor treatment): Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (Hb) ≥85g/L;

  •Liver function: Total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT) ≤3×ULN; Spread to the liver or liver cancer patient: 5 or less x ULN; Aspartate aminotransferase (AST) or less 3 x ULN; Spread to the liver or liver cancer patient: 5 or less x ULN;

  •Renal function: Creatinine (Cr) or less 1.5 x ULN; Creatinine clearance (Ccr) (calculated only when creatinine > 1.5× ULN) ≥50ml/min (calculated according to Cockcroft-Gault formula);

  •Blood coagulation function: Activated partial thromboplastin time (APTT) ≤1.5×ULN; International normalized ratio (INR) ≤1.5×ULN;

  •Urinary protein: Urine routine /24 hours urine protein qualitative ≤1+; Or urine protein qualitative ≥2+, 24 hours urine protein < 1g;
* 9. Expected survival of at least 3 months.
* 10. Women of childbearing potential had to have a negative serum or urine pregnancy test within 7 days before the first dose. Fertile male or female patients voluntarily during the study period and at the end of the study drug within 30 days of using effective birth control methods, such as abstinence, the double protective screen type cuts, condoms, contraceptive method of oral or injected contraceptives, intrauterine device, etc. All female patients will be considered fertile unless the female patient has undergone natural menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnophorectomy, or radioactive ovarian irradiation).

Exclusion Criteria:

* 1. The adverse reactions of previous antineoplastic therapy have not recovered to CTCAE 5.0 grade ≤1 (except for toxicities without safety risks judged by investigators, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stable with hormone replacement therapy);
* 2. Clinically symptomatic parenchymal or leptomeningeal metastases that were judged by the investigator to be ineligible for enrollment;
* 3. Within 4 weeks before delivery for the first time received chemotherapy, radiation therapy, biological therapy and endocrine therapy, immune therapy, such as antitumor drugs, with the exception of the following situations:

  * Nitrosourea or mitomycin C within 6 weeks before first use of study drug;
  * Oral fluorouracils and small-molecule targeted agents are administered 2 weeks before first use of the study drug or within the five half-lives of the drug, whichever is longer;
  * Have antitumor indications for the study of the first use of drugs of traditional Chinese medicines before 2 weeks;
* 4. Received other unlisted investigational drugs or treatments within 4 weeks before the first dose;
* 5. Previously received EP4 inhibitor (e.g. AN0025(E7046),LY3127760,ONO-4578) for anti-tumor treatment;
* 6. Major organ surgery (excluding needle biopsy) within 4 weeks before the first dose of medication or requiring elective surgery during the trial;
* 7. Uncontrolled malignant pleural, ascites, or pericardial effusion that was judged by the investigator to be ineligible for enrollment;
* 8. Unable to oral drug swallowing, or by the researchers determine the condition of the seriously affect the gastrointestinal tract absorption, including but not limited to, such as inflammatory bowel disease (crohn's disease and ulcerative colitis, for example), or malabsorption syndrome, or chronic diarrhea;
* 9. Patients who received a potent inducer or inhibitor of CYP3A4 within 1 week before the first dose or who required continued treatment with these drugs during the study;
* 10.Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases, or unresected tumor with active bleeding, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigator;
* 11.Thromboembolic events (including stroke events and/or transient ischemic attack) occurred within 12 months before the first dose of medication;
* 12.Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before the first dose of medication; Congestive heart failure with New York Heart Association (NYHA) grade ≥2; Left ventricular ejection fraction (LVEF) <50%; A history of primary cardiomyopathy, clinically significant prolongation of the QTc interval, or a screening QTc interval >470ms in women and >450ms in men;
* 13.Patients with active or previous autoimmune diseases with potential recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), excluding patients with clinically stable autoimmune thyroid diseases and type I diabetes mellitus;
* 14.Prior immunotherapy with grade ≥3 irAE or grade ≥2 immune-related myocarditis;
* 15.Researchers to determine the clinical significance of 3 or more electrolyte abnormalities
* 16.Patients with active infection requiring antiinfective treatment or unexplained fever (body temperature >38.5 ° C) during screening or before the first dose of medication;
* 17.Patients with active pulmonary tuberculosis (TB) who were receiving anti-TB treatment or had received anti-TB treatment within 1 year before the first dose; Known human immunodeficiency virus (HIV) infection; Patients with a history of hepatitis B were in the stage of active infection (HBsAg positive and HBV-DNA > the detection limit of the research center); Patients with a history of hepatitis C were in the active infection stage, defined as positive HCV antibody test and detectable HCV RNA;
* 18.Women who are pregnant (positive pregnancy test within 14 days before medication) or are breastfeeding
* 19.Patients with known alcohol or drug dependence;
* 20.Patients judged by the investigator that may not be able to comply with all study procedures;
* 21.Any other disease, metabolic abnormality, abnormal physical examinations or laboratory abnormality with significant clinical significance. Investigator reasonably suspects that the patient has a disease or state that is not suitable for using of the study drug, or will affect interpretation of study results, or put the patient at high risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 24 days after the initial drug administration
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0)
Maximum tolerated dose | Up to 24 days after the initial drug administration
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Recommended Dose for Phase II Clinical Studies (RP2D) | Up to 24 days after the initial drug administration
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of YY001.

SECONDARY OUTCOMES:
Duration of Response(DoR) | Up to approximately 24 months
  The time from the patient's first objective response to the patient's disease recurrence, progression, or death.
Overall Survival (OS) | Up to approximately 24 months
  The time from start date of study drug to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No